CLINICAL TRIAL: NCT06836843
Title: Evaluation of Maternal and Neonatal Outcomes Among Lebanese Women Conceived Through Assisted Reproductive Technology
Brief Title: Evaluation of Maternal and Neonatal Outcomes in Women Are Conceived Through Assisted Reproductive Technology Compared to Other Fertility Treatments and Naturally Conceived Women: It is a Retrospective Cohort Study Conducted Over a 5-year Period At a Fertility Center in a Lebanese Hospital
Acronym: non
Status: Active, not recruiting | Type: Observational
Sponsor: Lebanese University (Other)
Collaborators: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Reva Assem Mosleh, Principal Investigator, Lebanese University
Other Study IDs: BIO-2023-0200
Record Dates: First submitted 2024-12-10; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Preterm Birth; Gestational Diabetes Mellitus (GDM); Gestational Hypertension
Keywords: In vitro fertilization; IVF; Assisted reproductive technology; ART; neonatal outcome; neonatal complication; maternal outcome; maternal complication; pregnancy outcome; pregnancy complication; Intracytoplasmic sperm injection; spontaneous conception; fertility treatment; fertility management
MeSH Terms: conditions — Premature Birth; Diabetes, Gestational; Hypertension, Pregnancy-Induced; Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Exposed Group: The exposed group is subdivided into:
  Group one (Assisted Reproductive Technology group): pregnancies conceived via either in-vitro fertilization (IVF) with or without intracytoplasmic sperm injection (ICSI) with or without assisted hatching (AH) with or without pre-implantation genetic testing (PGT).
  Group two (Non-Assisted Reproductive Technology Group): pregnancies conceived through ovulation induction (OI) and/or intrauterine insemination (IUI) and/or corrective gynecological surgery.
  Interventions: Other: Since this is an observational study rather than an interventional study, the exposure type refers to all potential factors influencing pregnancy both before and during pregnancy
- Non-exposed Group: Spontaneous pregnancies, defined as pregnancies resulting from natural conception.
  Interventions: Other: Since this is an observational study rather than an interventional study, the exposure type refers to all potential factors influencing pregnancy both before and during pregnancy

INTERVENTIONS:
Other: Since this is an observational study rather than an interventional study, the exposure type refers to all potential factors influencing pregnancy both before and during pregnancy — Since this is an observational study rather than an interventional study or clinical trial, the exposure type refers to all potential factors influencing pregnancy both before conception and during pregnancy. These exposures include:
  Lifestyle habits: Such as obesity, smoking and alcohol use before and during pregnancy.
  Sociodemographic factors: Such as age, residence, medical insurance. Medications: Any prescription, over-the-counter, or herbal medications used before or during pregnancy.
  Past medical history: Pre-existing medical conditions or illnesses, such as hypertension, diabetes, or autoimmune diseases, that could affect pregnancy.
  Past surgical history: Previous surgeries, especially those related to the reproductive system or any that may impact pregnancy outcomes.
  Previous pregnancies: Information about past pregnancies, including the number of full-term and preterm births, complications, and outcomes.
  Abortions: Any history of miscarriages

SUMMARY:
Background: The number of couples experiencing difficulties conceiving and seeking treatment for infertility has increased dramatically over time. Treatment options for infertility have evolved significantly over the past four decades, expanding to include assisted reproductive technologies (ART). However, the impact of ART on pregnancy outcomes remains unclear. Studies have shown that ART pregnancies are associated with a higher risk of maternal and neonatal adverse outcomes compared to those resulting from spontaneous conception. To this date, no comprehensive studies have been conducted in Lebanon to assess this association. Therefore, it is crucial to evaluate whether Lebanese women who conceive via ART are at higher risk for maternal and birth-related complications.

Objective: The aim of this study is to evaluate maternal and neonatal outcomes among women who conceived through assisted reproductive technology (ART), compared to those who conceived via other fertility treatments or naturally, at Dr. Ghazeeri's clinic at the American University of Beirut Medical Center.

Methods: Investigators propose to conduct an observational retrospective cohort study involving all pregnant women treated by Dr. Ghazeeri who delivered at the American University of Beirut Medical Center between 2018 and 2023. Pregnancies exposed to assisted reproductive technology (ART) or other fertility treatments will be matched to a group of spontaneous pregnancies based on propensity scores. The study has been initiated following approval from the Institutional Review Board (IRB) at the American University of Beirut Medical Center. Data analysis will be performed using SPSS version 26.

Expected Results: If no associations are found between ART or other fertility treatments and an increased risk of maternal and neonatal outcomes, the results will provide reassurance for mothers seeking these treatments. However, if associations are identified, policymakers will need to establish comprehensive regulations outlining the appropriate use of these technologies. Additionally, these findings would lay the groundwork for obstetricians to implement closer monitoring and more careful management during pregnancy.

DETAILED DESCRIPTION:
i. Study Design Investigators propose to conduct an observational retrospective cohort study on all pregnant women who delivered at Dr. Gahzeeri's clinic at the American University of Beirut Medical Center between 2018 and 2023. Investigators have obtained approval from the Institutional Review Board (IRB) at AUB, which is valid until August 2025.

ii. Sample Size: As this is a retrospective cohort study, the sample size will be determined by the number of participants who meet the inclusion criteria.

iii. Population The patient characteristics will be extracted from the Epic electronic health record system at the hospital. Pregnancies exposed to ART or other fertility treatments will be matched to spontaneous pregnancies based on propensity scores

In this study, the subjects will be divided into two groups:

1. Exposed group:

   * Group One (ART group): pregnancies conceived via either IVF/ICSI and/or Assisted hatching (AH) and/or Pre-implantation genetic testing (PGT).
   * Group one will also be subdivided into fresh embryo transfer (ET) and frozen embryo transfer (FET) subgroups based on the type of embryo transfer method used.
   * Group Two (Non-ART group): pregnancies conceived through ovulation induction (OI) and/or intrauterine insemination (IUI) and/or corrective gynecological surgery.
2. Non-exposed group: spontaneous pregnancies, defined as pregnancies resulting from natural conception.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant ladies of Lebanese Nationality only who delivered at the American University of Beirut Medical Center (AUB-MC) between Nov 2018- Nov 2023
* Pregnancies that were delivered at least 20 weeks of gestation (≥ 20 weeks)
* All pregnant women who are in procreation age (20-50 years old)
* For pregnant women by ART: only if ART is done at the AUB-MC
* Subject's file being accessible for all the three trimesters
* Subjects being followed up until delivery only at the AUB-MC
* Subjects whom their baby or babies' records are available (it could be multiples)

Exclusion Criteria:

* Subjects who started their follow-up after the 1st trimester (missing data before 12 weeks).
* All subjects with history of severe chronic conditions before gestation such as, pre-existing cancer, heart diseases (coronary artery disease, arrhythmia, cardiac defects, ischemic stroke, venous thromboembolism, liver disease and/or kidney disease, history of nervous system disorders (seizures, depression).
* Subjects who undergone ART elsewhere
* Subjects who lost to follow up during their pregnancies (missing data)
* Moms who delivered outside the AUBMC hospital

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The eligibility for participation in this study is restricted to individuals who identify as female and are currently pregnant.
Study Population: It is an observational retrospective cohort study on all pregnant women who delivered at the American University of Beirut Medical Center between 2018 and 2023. The patient characteristics will be extracted from the Epic electronic health record system at the hospital. Pregnancies exposed to ART or other fertility treatments will be matched to spontaneous pregnancies based on propensity scores.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of Pregnant Women with Gestational Diabetes Mellitus (GDM) in the Exposed Group versus Non-Exposed Group | 24-28 weeks of gestation
  GDM will be diagnosed using standardized glucose screening tests; Oral Glucose Tolerance Test (OGTT) between 24 and 28 weeks of gestation.
  One-hour OGTT (after drinking a 50g glucose solution):
  Different cut-off thresholds are used for the 50-g glucose tolerance screening to be considered an abnormal result, including ≥130 mg/dL , ≥135 mg/dL, and ≥140 mg/dL.
  * Possible Gestational Diabetes (possible diagnosis if ≥140 mg/dL); and here the patient requires a confirmatory diagnosis which is the three-hours OGTT (after drinking 100g glucose solution):
  * Normal <140 mg/dL
  * Gestational Diabetes ≥140 mg/dL
Percentage of Pregnant Women with Gestational Hypertension in the Exposed Group versus the Non-Exposed Group | from 20 weeks + 1 day to 40 weeks of gestation
  Gestational hypertension is confirmed when blood pressure greater than or equal to 140mmHg systolic or 90mmHg diastolic on 2 separate occasions at least 4 hours apart after 20 weeks of pregnancy when previous blood pressure was normal
Percentage of Babies Born Preterm to Women in the Exposed Group versus Non-Exposed Group | Before 37 weeks of gestation
  Preterm is defined as babies born alive before 37 weeks of pregnancy are completed.
Percentage of Babies Born Small for Gestational Age to Women in the Exposed Group versus Non-Exposed Group | day one of birth
  Infants with a birth weight below the 10th percentile for their gestational age.
Percentage of Babies Born Large for Gestational Age to Women in the Exposed Group versus Non-Exposed Group | day one of birth
  Infants with a birth weight above the 90th percentile for their gestational age

SECONDARY OUTCOMES:
Percentage of Pregnant Women with Polyhydramnios in the Exposed Group versus Non-Exposed Group | During 40 weeks of gestation
  Polyhydramnios is usually defined as an amniotic fluid index (AFI) of more than 24 cm or a single pocket of fluid at least 8 cm in depth that results in an amniotic fluid volume of more than 2000 ml.
Percentage of Pregnant Women with Oligohydramnios in the Exposed Group versus Non-Exposed Group | During 40 weeks of gestation
  It is defined as an amniotic fluid index (AFI) less than 7 cm or the absence of a fluid pocket 2-3 cm in depth

OTHER OUTCOMES:
Percentage of Pregnant Women with Hypothyroidism in the Exposed Group versus Non-Exposed Group | During 40 weeks of gestation
  The diagnosis of hypothyroidism is made from the TSH value > 4.0 mIU/L.
Percentage of Pregnant Women with Hyperthyroidism in the Exposed Group versus Non-Exposed Group | During 40 weeks of gestation
  The diagnosis of hyperthyroidism is made from the TSH value <0.1 mUI/L

CONTACTS AND LOCATIONS:
Overall Officials: Ghina Ghazeeri, Professor of OBGYN and REI, Principal Investigator — American University of Beirut Medical Center; Amal Al Hajje, PhD in Clinical Pharmacy, Study Director — Professor at the Lebanese University; Roula Ajrouche, PhD in Epidemiology, Study Director — Associate Professor at the Lebanese University
Locations (1):
- Lebanese University, Beirut, Hadath, Lebanon

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) shared will be fully de-identified. No personally identifiable information (PII) will be included in the dataset. All data will be anonymized to ensure participant privacy and confidentiality, in accordance with applicable privacy and ethical guidelines.
  The data collection sheet includes information on sociodemographic factors, past medical and surgical history, lifestyle habits, previous pregnancy details, medication use before and during pregnancy, assisted reproductive technology (ART) procedures (including type, year, embryo type, and ovulation induction medication), infertility history and its causes, as well as pregnancy-related and neonatal outcomes. Specifically, it captures details such as age, medical conditions, medications, mode of delivery, maternal complications (e.g., hypertension, diabetes, and others), and neonatal outcomes (e.g., APGAR score, birth weight, prematurity, and others).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Graham ME, Jelin A, Hoon AH Jr, Wilms Floet AM, Levey E, Graham EM. Assisted reproductive technology: Short- and long-term outcomes. Dev Med Child Neurol. 2023 Jan;65(1):38-49. doi: 10.1111/dmcn.15332. Epub 2022 Jul 18. PMID 35851656
- [Background] Vermey BG, Buchanan A, Chambers GM, Kolibianakis EM, Bosdou J, Chapman MG, Venetis CA. Are singleton pregnancies after assisted reproduction technology (ART) associated with a higher risk of placental anomalies compared with non-ART singleton pregnancies? A systematic review and meta-analysis. BJOG. 2019 Jan;126(2):209-218. doi: 10.1111/1471-0528.15227. Epub 2018 May 8. PMID 29740927
- [Background] Chih HJ, Elias FTS, Gaudet L, Velez MP. Assisted reproductive technology and hypertensive disorders of pregnancy: systematic review and meta-analyses. BMC Pregnancy Childbirth. 2021 Jun 28;21(1):449. doi: 10.1186/s12884-021-03938-8. PMID 34182957
- [Background] Bosdou JK, Anagnostis P, Goulis DG, Lainas GT, Tarlatzis BC, Grimbizis GF, Kolibianakis EM. Risk of gestational diabetes mellitus in women achieving singleton pregnancy spontaneously or after ART: a systematic review and meta-analysis. Hum Reprod Update. 2020 Jun 18;26(4):514-544. doi: 10.1093/humupd/dmaa011. PMID 32441298
- [Background] Qin J, Liu X, Sheng X, Wang H, Gao S. Assisted reproductive technology and the risk of pregnancy-related complications and adverse pregnancy outcomes in singleton pregnancies: a meta-analysis of cohort studies. Fertil Steril. 2016 Jan;105(1):73-85.e1-6. doi: 10.1016/j.fertnstert.2015.09.007. Epub 2015 Oct 9. PMID 26453266